CLINICAL TRIAL: NCT07329946
Title: Erdosteine Effect on Oxidative Stress, Inflammatory Response and Immune Modulation in Patients With COPD. A Single Center, Open Label, Double Arm, Controlled, 4-week, Explorative, ex Vivo Study."
Brief Title: Immuno-inflammatory Response of Erdosteine in COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pierachille Santus, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Pierachille Santus, MD, PhD, Professor, University of Milan
Organization: University of Milan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400.141CRC
Record Dates: First submitted 2025-12-10; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: COPD
Keywords: COPD; ERDOSTEINE
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — erdosteine; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A - Erdosteine treatment (Experimental): Patients will be randomized to receive Erdosteine [Esteclin®] 300 mg, 1 tablet twice daily for 30 days
  Interventions: Drug: Erdosteine; Drug: Standard of Care (SOC)
- ARM B - Standard of care (Placebo Comparator): Patients will be randomized to receive current standard inhalation therapy in use
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: Erdosteine — Erdosteine tablets 300 mg, 1 tablet orally every 12 hours (twice daily) for 30 days
  Other Names: Esteclin
  Arms: ARM A - Erdosteine treatment
Drug: Standard of Care (SOC) — Long acting beta-2 agonists and Long acting muscarinic antagonists in association (LABA/LAMA) with or without inhaled corticosteroids (LABA/LAMA/ICS) depending on the chronic inhaled home treatment. Dosage and posology will change depending on the molecules and the devices (once daily in case of umeclidinium bromide/vilanterol 55/22 mcg or fluticasone/umeclidinium bromide/vilanterol 92/55/22 or twice daily in case of budesonide/formoterol/glycopyrronium 160/7.2/4.8 mcg and beclometasone/formoterol/glycopyrronium 87/5/9 mcg)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) remains a major contributor to global morbidity and mortality, exposing healthcare systems to a significant economical and social load. Indeed, acute severe COPD exacerbations are the events that contribute most to the overall disease burden. Current management strategies are aimed at maximizing symptom-free periods, reduce hospitalizations, improve exercise tolerance, overall health status, and quality of life. Key pathophysiological mechanisms involved in COPD exacerbations (defined as acute worsening of respiratory symptoms) include oxidative stress, acute on chronic inflammation, and mucus hypersecretion. Agents with antioxidant, anti-inflammatory, and mucolytic properties can help reduce exacerbation frequency. Erdosteine is a new-generation mucoactive molecule developed to overcome the limitations associated with traditional mucolytics. In fact, in addition to its mucolytic effects, erdosteine exhibits antioxidant and anti-inflammatory activities and may reduce bacterial adhesion to airway surfaces - features that may be beneficial in the prevention and management of exacerbations. Preliminary clinical findings (EQUALIFE and RESTORE studies) suggest that erdosteine, in add-on to chronic inhaled therapy, can reduce exacerbation rates, shorten hospital stay, and improve health-related quality of life in patients with COPD. However, studies that have investigated the pathobiological mechanisms behind such clinical effects are lacking.

The present study was constructed in order to investigate the mechanism of action of erdosteine on inflammation, oxidative stress pathways and immune response in patients with COPD. The secondary objectives of the study are to evaluate the effect of erdosteine on lung function tests in patients with COPD; to explore the effect of erdosteine on respiratory and COPD-related symptoms in patients with COPD; to assess the effect of erdosteine on exercise tolerance in patients with COPD. In order to do so, the investigator designed a pragmatic, low intervention, two-arms, monocenter, open-label, prospective, randomized, controlled trial, set in clinical practice. A total of 30 patients will be randomized by means of a 1:1 random allocation.

The active group (15 patients) will be assigned to Treatment Arm A (Erdosteine [Esteclin®] 300 mg, 1 tablet twice daily for 30 days), while the control group (15 patients) will be assigned to Treatment Arm B (Standard of Care - current standard inhalation therapy in use).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years
2. A confirmed COPD diagnosis at least 12 months prior to enrollment
3. Stable clinical conditions, defined as no exacerbations or respiratory infections of any severity in the last 3 months before enrollment
4. Moderate to Severe airflow obstruction (FEV1 30-80 %predicted post bronchodilation.
5. No hospitalizations for any cause in the 3 months prior to enrollment
6. Ability to perform repeatable pulmonary function tests
7. Chronic inhaled therapy with LAMA/LABA or LAMA/LABA/ICS with no changes in dosage in the last 3 before enrollment

Exclusion Criteria:

1. NYHA class III and IV heart failure
2. Unstable arrythmia
3. Active malignancy (solid or blood)
4. Chronic treatment with systemic corticosteroids or immunosuppressants
5. Immune depression
6. Known hypersensitivity to erdosteine
7. Pregnancy or breastfeeding

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in transcriptomics of pro-inflammatory and anti-inflammatory cytokines in COPD patients exposed to erdosteine. | 4 weeks
  Peripheral blood will be analyzed for immunological profiling in patients treated with standard of care only and patients also exposed to Erdosteine at baseline and after 4 weeks of treatment. Cytokine/chemokine profiles will be quantified in cell culture supernatants using the Bio-Plex Pro Human Cytokine 27-plex Assay. RNA extraction from whole blood will be performed to identify expression levels of molecules involved in immune response: CARD6, CASP1, CASP4, CCL2, HLA-A, IFITM1, IFNA1, IFNAR1, IL1β, IL6, IL8, IL10, IL17, IL18, IL22, ISG20, TGF-β, NLRP3, NLRP4, VCAM1. Betaactin (ACTB) and glyceraldeyde-3-phosphate dehydrogenase (GAPDH) will be used as housekeeping genes. The results for the gene expression analyses will be presented as the average of the relative expression units (%) to an internal reference sample and normalized to the housekeeping genes GAPDH and ACTB.
Changes in transcriptomics of oxidative stress signaling pathways in COPD patients exposed to erdosteine. | 4 weeks
  Peripheral blood will be analyzed for oxidative stress profiling in patients treated with standard of care only and patients also exposed to Erdosteine at baseline and after 4 weeks of treatment. Oxidative stress will be quantified in cell culture supernatants using the Bio-Plex Pro Human Cytokine 27-plex Assay. RNA extraction from whole blood will be performed to identify expression levels of molecules involved in oxidative stress: APOE, CAT, DUSP1, GPX2, GPX3, MPO, NOS2, NOX4, NUDT1, SOD2. Betaactin (ACTB) and glyceraldeyde-3-phosphate dehydrogenase (GAPDH) will be used as housekeeping genes. The results for the gene expression analyses will be presented as the average of the relative expression units (%) to an internal reference sample and normalized to the housekeeping genes GAPDH and ACTB.

SECONDARY OUTCOMES:
To assess the effect of erdosteine on mMRC dyspnea scale in patients with COPD | 4 weeks
  Patiens will undergo the Modified British Medical Research Council Questionnaire (mMRC) at baseline and after 4 weeks of treatment with erdosteine or placebo.
  Modified British Medical Research Council Questionnaire (mMRC) assesses the patient's degree of chronic dyspnea with a score ranging from 0 (no dyspnea) to 4 (too much dyspnea to leave the house). The results will be expressed as absolute and relative difference in dyspnea score.
To assess the effect of erdosteine on distance covered during the six minute walk test in patients with COPD | 4 weeks
  Patiens will undergo the Six Minutes Walk Test (6MWT) at study enrolment and after 4 weeks of treatment with erdosteine or placebo.
  The 6MWT will be conducted according to the 2002 American Thoracic Society (ATS) statement. For patients requiring exertional oxygen therapy, the test will be performed with supplemental oxygen. Patients will be asked to walk for 6 minutes on a flat surface, wearing a pulse oximeter. Before starting, the following parameters will be recorded: perceived dyspnoea level using the Borg scale (0-10 score), peripheral oxygen saturation (SpO2), heart rate (beats/min), and respiratory rate (breaths/min). The same parameters will be measured again at the end of the test. The distance walked, and any exercise-induced desaturation (SpO2 drop ≥4 points) will also be noted. The distance covered at the 6MWT will be measured in meters, and results will be expressed as absolute and relative difference from baseline.
To assess the effect of erdosteine on CAT (COPD assessment test) in patients with COPD | 4 weeks
  Patiens will undergo the CAT (COPD assessment test) at baseline and after 4 weeks of treatment with erdosteine or placebo.
  COPD assessment test (CAT) aims to assess the impact of COPD on health status through a patient-completed questionnaire consisting of 8 items, each scored from 0 to 5. The total score ranges from 0 to 40, with higher scores indicating a greater impact of the disease on the patient's quality of life. The results will be expressed as absolute and relative difference in CAT total score.

OTHER OUTCOMES:
To evaluate the effect of erdosteine on dynamic lung volumes in patients with COPD | 4 weeks
  Dynamic lung volumes, will be measured using a constant-volume body plethysmograph at study enrolment and after 4 weeks of treatment with erdosteine or placebo.
  The following volumes will be measured: forced expiratory volume in first second (FEV₁), forced vital capacity (FVC), slow VC, forced mid-expiratory flow at 25 and 75% of FVC (FEF25-75), expiratory reserve volume (ERV). The results will be expressed as absolute (liters) and % predicted value, and measured as absolute and relative difference from baseline.
To assess the effect of erdosteine on static volumes in patients with COPD | 4 weeks
  Static lung volumes will be measured using a constant-volume body plethysmograph according to current recommendations (Wanger et al. Eur Respir J 2005) at baseline and after 4 weeks of treatment with erdosteine or placebo.
  Patients will be instructed to breathe in seated position, wearing a nose clip, while connected to a pneumotachograph, with closed cabin. The following volumes will be measured: residual volume (RV), total lung capacity (TLC), RV/TLC and intrathoracic gas volume (ITGV). ITGV will be measured close to the end-expiratory lung volume during quiet breathing to obtain functional residual capacity (FRC). The results will be expressed as absolute (liters) and % predicted value, and measured as absolute and relative difference from baseline.
To evaluate the effect of erdosteine on lung diffusion capacity in patients with COPD | 4 weeks
  Lung diffusion capacity for carbon monoxide (DLCO) will be measured using a constant-volume body plethysmograph at study enrolment and after 4 weeks of treatment with erdosteine or placebo.
  DLCO, transfer factor (KCO), and alveolar volume (VA) will be measured using the single-breath technique. VA will be assessed by means of the inert gas dilution technique. The DLCO value will be corrected based on the most recent available hemoglobin value. The results will be expressed as absolute (mmol x min-1 kPa-1 for DLCO, mmol x min-1 kPa-1 1-1 for KCO, and liters for VA) and % predicted value, and measured as absolute and relative difference from baseline.
To evaluate the effect of erdosteine on specific airway resistances in patients with COPD | 4 weeks
  Specific airway resistances (sRAW) will be measured using a constant-volume body plethysmograph according to current recommendations (Wanger et al. Eur Respir J 2005) at baseline and after 4 weeks of treatment with erdosteine or placebo. Patients will be instructed to breathe tidally in seated position, wearing a nose clip, while connected to a pneumotachograph, with closed cabin. The results will be expressed as absolute (kPa x s) and % predicted value, and measured as absolute and relative difference from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided